CLINICAL TRIAL: NCT01677364
Title: ELECTIVE INDUCTION OF LABOUR VS SPONTANEOUS LABOUR IN WOMEN WITH HEART DISEASE - A PROSPECTIVE RANDOMIZED CONTROLLED TRIAL
Brief Title: Elective Induction vs Spontaneous Labour in Patients With Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Yogita Dogra, Dr.Yogita Dogra, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7862/PG/2Trg/08
Record Dates: First submitted 2012-08-26; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Heart; Disease,Complicating Pregnancy, Pre-existing
Keywords: induction of labour; heart disease patients
MeSH Terms: conditions — Disease; Pregnancy Complications | interventions — Oxytocin

ARMS (2):
- induction of labour (Active Comparator): drug- infusion of 30U oxytocin diluted in 500ml normal saline given at rate of 3mU/min and subsequently dose increased 3mU/min every 45 min
  Interventions: Drug: Oxytocin
- Spontaneous Labour (No Intervention): patients were allowed to go into spontaneous labour

INTERVENTIONS:
Drug: Oxytocin — Arm - Induction of labour
  Arms: induction of labour

SUMMARY:
Fifty pregnant patients with acquired and congenital heart disease between 38-41 weeks were randomised into elective induction and spontaneous labour groups only after bishop score was equal to or more than 6.It was concluded that induction of labour with oxytocin is a relatively safe procedure in women with low risk heart disease with NYHA class I and II. It resulted in a similar caesarean delivery rate and was not associated with more maternal and neonatal complications.

DETAILED DESCRIPTION:
Induction of labour was done with oxytocin. An infusion of 30U oxytocin diluted in 500ml normal saline was prepared and given through infusion pump at initial rate of 3mU/min. Subsequently dose was increased 3mU/min every 45 min till adequate uterine contractions were established.

Epidural analgesia was provided wherever feasible or Injection Morphine 2-5mg was given intravenously for pain relief.

ELIGIBILITY:
Inclusion Criteria:

* NYHA class I-II
* cephalic presentation
* singleton gestation

Exclusion Criteria:

* previous cesarean section,
* Primary pulmonary hypertension,
* Eisenmenger syndrome,
* Marfan syndrome,
* Left heart obstruction,
* Prior cardiac event or arrhythmia,
* Malformed fetus,
* Severe anemia (<7g/dl),
* Intrauterine fetal death,
* other obstetrical indications for induction of labour
* patients on anticoagulation.

Ages: 19 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Duration of labour | at the time of delivery
Rate of caesarean section | at the time of delivery
  mode of delivery and rate of caesarean section with indication
Number of patients with delivery during workday hours | at the time of delivery

SECONDARY OUTCOMES:
number of patients with maternal complications | day 5
  maternal complications include postpartum hemorrhage, infection, cardiac complications and number of maternal deaths
number of patients with adverse neonatal outcome | day 5
  apgar score number of admissions to neonatal intensive care unit number of neonatal deaths

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India